CLINICAL TRIAL: NCT07086261
Title: The Effectiveness of Using Spaced Retrieval Training to Improve The Drinking Problem Behavior of Elderly People With Dementia During The Care of Day Care Centers in Taoyuan, Taiwan
Brief Title: Using SRT to Improve The Drinking Problem Behavior of Elderly People With Dementia During The Care of Day Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Wu Chia Jung, Principal Investigator, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202501EM036
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer's Disease (AD)
Keywords: Alzheimer's Disease; Spaced Retrieval Training; Water, drinking; Memory; Fluid intake

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Intervention of timed retrieval training program to implement relevant water drinking training
  Interventions: Other: Spaced Retrieval Training
- Drink water as usual (No Intervention)

INTERVENTIONS:
Other: Spaced Retrieval Training — This study adopted a quasi-experimental research design with two groups of pre- and post-tests. The sample was recruited by convenient sampling. The experimental group used the time extraction training program to intervene and perform relevant water drinking training, 40 minutes each time, 3 times a week, for a total of 8 weeks of intervention measures, while the control group used routine care for general water drinking. Both groups collected pre-test data before the time extraction training intervention program activities in the first week, and conducted post-test data tracking and analysis in the 4th and 8th weeks after the intervention activities.
  Arms: Experimental Group

SUMMARY:
Objective: To explore the effects of intermittent retrieval training on cognitive function, daily water intake, body weight, total body water, drinking problem behaviors in day care centers, and caregiver distress in day care centers for elderly people with dementia.

Methods: This study adopted a quasi-experimental research design with two groups of pre- and post-tests. The sample was recruited by convenient sampling. The experimental group was intervened with the intermittent retrieval training program to perform relevant drinking training, 40 minutes each time, 3 times a week, for a total of 8 weeks of intervention measures, while the control group was carried out with routine care for general drinking. Both groups collected pre-test data before the intermittent retrieval training intervention program in the first week, and conducted post-test data tracking and analysis in the 4th and 8th weeks after the intervention activities. The research tools included basic attribute data sheet, Chinese version of cognitive ability screening test (CASI), daily water intake, average daily water intake and drinking problem behaviors in the past week, body fat scale for measuring weight and total body water content, and day care center caregiver burden assessment scale. It is expected that this research intervention measure can improve the behavior of elderly people with dementia to drink water independently.

DETAILED DESCRIPTION:
Background: Elderly people with dementia have impaired semantic and episodic memory, which significantly affects the difficulties of caregivers in day care centers and the burden of primary caregivers. During their internship in nursing care for the elderly at graduate school, researchers found that many elderly people with dementia have drinking problems. Some elderly people did not drink enough water, which caused their skin to be dry and flaky. They also forgot to replenish water after many dynamic activities in the course, which caused them to sweat too much. Many female elderly people also suffered from urinary tract infections. Therefore, if a training program can be designed for each elderly person to use time retrieval training as drinking behavior training, it will not only improve the memory of elderly people with mild cognitive impairment and dementia, but also enhance the training of the elderly in daily life functions, so as to increase the daily water intake to improve the physical burden and the occurrence of diseases and the burden on day care centers or family caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Elderly people with dementia aged 65 years or above who are receiving care in day care centers.
* Clear consciousness and able to communicate in Mandarin and Taiwanese.
* Clinical Dementia Rating Scale (CDR) should be 1-2 points.
* Brain Health Test (BHT) should be less than 9 points.
* Pass the SRT training screening test, indicating that the trainer's name can be remembered for 20-30 seconds.
* Agree to participate in this study.

Exclusion Criteria:

* Patients diagnosed with severe cognitive impairment according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) after evaluation by psychiatrists.
* Patients with chronic heart disease and renal failure.
* Patients with upper and lower limb dysfunction.
* Patients with hearing impairment and dysphagia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive function (CASI) | 10-20minute
  Total number of questions: 25, The higher the score, the better, with a full score of 100, indicating better cognitive function. Taking high school graduates as an example, a score of 82 or more is considered normal, 78-81 is suspected of mild cognitive impairment, and less than 77 is considered suspected of dementia.
Daily water intake and Drinking Problem Behavior | From intervention to end of 8 weeks
  Calculate the water requirement of the elderly according to the recommended daily water requirement per person by multiplying 30 mL per kilogram of body weight (e.g., if the elderly weigh 60 kg, 60 kg × 30 ml = 1800 ml, 1800 ml/day). While the elderly are at the day care center, researchers and staff will monitor their water intake. When they return home from the center, researchers will give each person a 600ml bottle of mineral water (the bottle will be marked with the total amount of water the elderly need to drink in a day). Elderly people are asked to take it home, and family members are asked to help monitor the elderly's water intake at home. Family members are asked to deduct the amount of water they drink and record the remaining amount of water in the "Elderly Drinking Water Good Health Plan Water Drinking Registration Form"and"Daily Water Intake Registration Form for Elderly People"
Distress of caregivers in day care centers | From intervention to end of 8 weeks
  There are 10 questions in total, used in the questionnaire on the concerns of caregivers about drinking water problems of elderly people with dementia.The scale is a Likert scale with a 0-4 point scale, with a total of 40 points.The higher the score, the more trouble the caregiver has with the subject's drinking behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Taoyuan Branch, Taipei Veterans General Hospital., Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] Han JW, Son KL, Byun HJ, Ko JW, Kim K, Hong JW, Kim TH, Kim KW. Efficacy of the Ubiquitous Spaced Retrieval-based Memory Advancement and Rehabilitation Training (USMART) program among patients with mild cognitive impairment: a randomized controlled crossover trial. Alzheimers Res Ther. 2017 Jun 6;9(1):39. doi: 10.1186/s13195-017-0264-8. PMID 28587629
- [Background] Kao CC, Lin LC, Wu SC, Lin KN, Liu CK. Effectiveness of different memory training programs on improving hyperphagic behaviors of residents with dementia: a longitudinal single-blind study. Clin Interv Aging. 2016 May 23;11:707-20. doi: 10.2147/CIA.S102027. eCollection 2016. PMID 27307717
- [Background] Bunn DK, Abdelhamid A, Copley M, Cowap V, Dickinson A, Howe A, Killett A, Poland F, Potter JF, Richardson K, Smithard D, Fox C, Hooper L. Effectiveness of interventions to indirectly support food and drink intake in people with dementia: Eating and Drinking Well IN dementiA (EDWINA) systematic review. BMC Geriatr. 2016 May 4;16:89. doi: 10.1186/s12877-016-0256-8. PMID 27142469
- [Background] Wu HS, Lin LC, Wu SC, Lin KN, Liu HC. The effectiveness of spaced retrieval combined with Montessori-based activities in improving the eating ability of residents with dementia. J Adv Nurs. 2014 Aug;70(8):1891-901. doi: 10.1111/jan.12352. Epub 2014 Jan 20. PMID 24444172
- [Background] Wu HS, Lin LC, Su SC, Wu SC. The effects of spaced retrieval combined with errorless learning in institutionalized elders with dementia: recall performance, cognitive status, and food intake. Alzheimer Dis Assoc Disord. 2014 Oct-Dec;28(4):333-9. doi: 10.1097/WAD.0000000000000028. PMID 24632986